CLINICAL TRIAL: NCT06778057
Title: Clinical Performance of Three Daily Disposable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6595
Record Dates: First submitted 2024-12-27; First posted 2025-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Test Lens 1/Test Lens 2/Test Lens 3 (Experimental): Eligible subjects will be randomized into the Test Lens 1/Test Lens 2/Test Lens 3 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3
- Test Lens 1/Test Lens 3/Test Lens 2 (Experimental): Eligible subjects will be randomized into the Test Lens 1/Test Lens 3/Test Lens 2 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3
- Test Lens 2/Test Lens 1/Test Lens 3 (Experimental): Eligible subjects will be randomized into the Test Lens 2/Test Lens 1/Test Lens 3 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3
- Test Lens 2/Test Lens 3/Test Lens 1 (Experimental): Eligible subjects will be randomized into the Test Lens 2/Test Lens 3/Test Lens 1 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3
- Test Lens 3/Test Lens 1/Test Lens 2 (Experimental): Eligible subjects will be randomized into the Test Lens 3/Test Lens 1/Test Lens 2 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3
- Test Lens 3/Test Lens 2/Test Lens 1 (Experimental): Eligible subjects will be randomized into the Test Lens 3/Test Lens 2/Test Lens 1 sequence, to wear each lens for up to 10 hours each.
  Interventions: Device: Test Lens 1; Device: Test Lens 2; Device: Test Lens 3

INTERVENTIONS:
Device: Test Lens 1 — Acuvue® Oasys MAX 1-Day daily disposable contact lenses
Device: Test Lens 2 — Dailies Total 1 daily disposable contact lenses
Device: Test Lens 3 — Clariti 1-Day daily disposable contact lenses

SUMMARY:
This is a subject-masked, randomized, prospective, bilateral, 3x3 crossover dispensing clinical investigation to assess the clinical performance of a new lens type comparison.

ELIGIBILITY:
Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 40 (inclusive) years of age at the time of screening.
4. By self-report, they typically use digital devices for a minimum of 4 hours per day, 5 days per week.
5. In a pre-study screening assessment, they must have a CVS-Q score of 6 or greater.
6. Agree not to participate in other clinical research while enrolled on this study.
7. Own a wearable pair of spectacles, if needed, for distance vision correction (by self-report).
8. By self-report, habitually wear silicone hydrogel soft contact lenses in both eyes in a daily reusable or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 8 hours of wear per day, for at least 4 days per week over the past 4 weeks.
9. Attain a best-corrected logMAR distance visual acuity of at least 0.20 in each eye.
10. Have spherical contact lens prescription in the range -1.00 to -6.00 DS (based on the calculated ocular refraction) in each eye.
11. Have up to a maximum of 1.00 DC of refractive astigmatism (based on the calculated ocular refraction) in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

1. Be currently pregnant or lactating.
2. By self-report, have any systemic disease (e.g., Sjögren's Syndrome), allergies, infectious disease (e.g. hepatitis, tuberculosis), contagious immunosuppressive diseases (e.g., HIV), autoimmune disease (e.g., rheumatoid arthritis), or other diseases, which in the opinion of the investigator is likely to interfere with contact lens wear and/or participation in the study or may pose a risk to study personnel.
3. Have an ocular disorder which would normally contraindicate contact lens wear.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing monovision or multifocal contact lenses.
6. Be currently wearing or have had worn Acuvue® Oasys 1-Day, Dailies® Total1, or Clariti 1-Day lenses during the last 3 months.
7. Have had cataract surgery.
8. Have had corneal refractive surgery.
9. Be using any topical medications such as eye drops or ointments.
10. Have a known hypersensitivity or allergic reaction to sodium fluorescein.
11. Use of systemic medications (e.g., chronic steroid use) that are known to interfere with contact lens wear. See section 9.1 for additional details regarding excluded systemic medications.
12. Participation in any contact lens or lens care product clinical trial within 2 weeks prior to study enrolment
13. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
14. Have clinically significant (grade 3 or higher on the Efron grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that in the opinion of the investigator would contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis).
15. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
16. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-12-29 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Lens Fit Acceptance | Follow-up assessments will be made approximately 8-10 hours after lens dispensing
  Lens Fit Acceptance: Lens fit acceptance will be assessed at dispensing and follow-up visits for each subject eye.
  An unacceptable fit is deemed by one or more of the following criteria:
  * limbal exposure at primary gaze or with extreme eye movement.
  * edge lift.
  * excessive movement with blink in primary gaze.
  * insufficient movement with blink in upgaze.
  * insufficient movement in push-up test.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester, Department of Optometry & Neuroscience, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu